CLINICAL TRIAL: NCT00488605
Title: H-9926-LCH III: Treatment Protocol of the Third International Study for Langerhans Cell Histiocytosis
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: This is a duplicate record and the sponsor has registered the study.
Sponsor: University of New Mexico (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-9926-LCH III
Record Dates: First submitted 2007-06-14; First posted 2007-06-20 (Estimated); Last update posted 2023-08-03 (Actual); Status verified 2023-08

CONDITIONS: Leukemia
MeSH Terms: conditions — Leukemia | interventions — Prednisone; Vinblastine; Leucovorin; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment Arm A (Active Comparator)
  Interventions: Drug: Prednisone, Vinblastin, 6-mercaptopuroine
- Treatment Arm B (Experimental)
  Interventions: Drug: Leucovorin, Methotrexate, Vinblastine, Prednisone

INTERVENTIONS:
Drug: Prednisone, Vinblastin, 6-mercaptopuroine — Initial Therapy:Prednisone- by mouth 3 times/day daily as a 4-week course, then gradually decreased over 2 more weeks. Vinblastine-IV (into a vein)1 day/week for 6 weeks. Patients w/o evidence of active disease at this time will proceed to continuation therapy. If disease is improved or unchanged, pts. will receive additional therapy with: Prednisone- 3 divided doses by mouth for 3 days every week, from week 7-12. Vinblastine- IV 1day/week for 6 more weeks. If the disease is gone or better after this additional therapy continuation will begin. Continuation Therapy: 6-MP:by mouth daily until the end of month 12. Prednisone in 3 doses daily day 1-5 every 3 weeks until the end of month 12. Vinblastine IV day 1 every 3 weeks until the end of month 12.
  Arms: Treatment Arm A
Drug: Leucovorin, Methotrexate, Vinblastine, Prednisone — Initial Therapy:Prednisone-by mouth 3x/day daily as a 4-week course then gradually decreased over 2 more weeks. Vinblastine- IV 1 day/week for 6 weeks. Methotrexate-a 24 hour IV infusion day 1 of weeks 1, 3, and 5, followed by leucovorin.The drug will be given by mouth. Pts w/o evidence of active disease at this time will proceed to continuation therapy. Pts whose disease is improved or unchanged will receive additional therapy w/:Prednisone- 3 divided doses, days 1-3 weekly from week 7-12. Vinblastine IV 1day/week for 6 more weeks. Methotrexate-a 24 hour IV infusion day 1 of week 7, 9, and 11, followed by leucovorin. If the disease is gone or better after this additional therapy continuation will begin. Continuation Therapy: 6-MP by mouth daily until the end of month 12. Prednisone- 3 doses daily days 1-5 every 3 weeks until the end of month 12. Vinblastine IV day 1 every 3 weeks until the end of month 12. Methotrexate by mouth once weekly until the end of month 12.
  Other Names: leukovorin rescue
  Arms: Treatment Arm B

SUMMARY:
LCH III is an international, multicentric, prospective clinical study comprised of:

* a randomized clinical trial for multisystem "RISK" patients and
* a randomized clinical trial for multisystem "LOW RISK" patients and
* a pilot study for patients with single system MFB and localized "SPECIAL SITES"

DETAILED DESCRIPTION:
Therapy for "LOW RISK" Patients:

The decision as to which research program you will be assigned will be made entirely by chance. The overall time of therapy will be 6 or 12 months as randomly assigned. The research program will be with the drugs Vinblastine and Prednisone.

Initial Therapy

1. Prednisone given by mouth three times a day daily as a four-week course, then gradually decreased over 2 more weeks.
2. Vinblastine will be given IV (into a vein) one day a week for 6 weeks.
3. Patients who have no evidence of active disease at this time will proceed to continuation therapy.

Patients whose disease response is stable, mixed or worse will receive additional therapy with:

1. Prednisone in 3 divided doses by mouth for 3 days every week, from week 7-12.
2. Vinblastine IV one day a week for 6 more weeks.

   * If the disease is gone or better after this additional therapy continuation will begin.

Continuation Therapy

1. Prednisone in 3 doses daily day 1-5 every 3 weeks until the end of month 6 or 12 from start of therapy, as randomized.
2. Vinblastine IV day 1 every 3 weeks until the end of month 6 or 12 from start of therapy, as randomized.

Therapy for "SPECIAL SITE" (Multi-focal Bone Involvement) Patients:

Treatment consists of an initial treatment of 6 weeks and a continuation treatment. A second course is given only to patients with progressive disease. The overall therapy time period is 6 months.

Initial Therapy 4. Prednisone given by mouth three times a day daily as a four-week course, then gradually decreased over 2 more weeks.

5. Vinblastine will be given IV (into a vein) one day a week for 6 weeks. 6. Patients who have no evidence of active disease at this time will proceed to continuation therapy.

Patients whose disease response is stable, mixed or worse will receive additional therapy with:

3. Prednisone in 3 divided doses days 1-3 weekly from week 7-12. 4. Vinblastine IV one day a week for 6 more weeks.

* If the disease is gone or better after this additional therapy continuation will begin.

Continuation Therapy 3. Prednisone in 3 doses daily day 1-5 every 3 weeks until the end of month 6. 4. Vinblastine IV day 1 every 3 weeks until the end of month 6.

Group 1 "RISK" patients:

The primary aim of the study is to compare the therapeutic efficacy of control arm A (PDN+VBL) with the experimental arm B (PDN+VBL+MTX). The primary endpoint is the proportion of non-responder in risk organs to the initial treatment.

Non-response to initial therapy is defined as:

• death within 12 weeks of initial treatment or

* progression (worse) in risk organs at week 6
* lack of response (=intermediate response or progression) in risk organs at week 12 as compared to the status of disease at week 6.

If the null hypothesis is true, the two randomized treatment arms are equally effective in terms of non-response. If the alternative hypotheses is true, there is a difference between the two randomized arms in terms of efficacy.

Group 2 "LOW RISK" patients:

The primary aim of the study is to compare the reactivation free survival rate in initial responders at week 6 with continuation treatment for 6 months (Arm LR 6) versus 12 months (Arm LR 12) in those patients without disease reactivation within the first 6 months.

If the null hypothesis is true, the reactivation rate of both randomized arms are equal. If the alternative hypothesis is true, there is a difference between the two arms in terms of reactivation frequency.

Therapy for "RISK" Patients:

Treatment A will consist of:

7. Initial Therapy 8. Prednisone given by mouth three times a day daily as a four-week course, then gradually decreased over 2 more weeks.

9. Vinblastine will be given IV (into a vein) one day a week for 6 weeks. 10. Patients who have no evidence of active disease at this time will proceed to continuation therapy.

Patients whose disease is improved or unchanged will receive additional therapy with:

5. Prednisone in 3 divided doses by mouth for 3 days every week, from week 7-12.

6. Vinblastine IV one day a week for 6 more weeks.

** If the disease is gone or better after this additional therapy continuation will begin.

Continuation Therapy:

5. 6-MP by mouth daily until the end of month 12. 6. Prednisone in 3 doses daily day 1-5 every 3 weeks until the end of month 12. 7. Vinblastine IV day 1 every 3 weeks until the end of month 12.

** Those patients whose disease didn't respond to the initial therapy by the 12th week will come off this study and proceed to other research programs.

Treatment B will consist of:

1. Initial Therapy
2. Prednisone given by mouth three times a day daily as a four-week course then gradually decreased over 2 more weeks.
3. Vinblastine will be given IV one day a week for 6 weeks.
4. Methotrexate given as a 24 hour IV infusion day 1 of weeks 1, 3, and 5, followed by leucovorin.
5. Leucovorin is a drug that will be given to help the body remove the methotrexate and decrease the possible side effects. (This is sometimes called a "leukovorin rescue". The drug will be given by mouth.)

   * Patients who have no evidence of active disease at this time will proceed to continuation therapy.

Patients whose disease is improved or unchanged will receive additional therapy with:

1. Prednisone in 3 divided doses, days 1-3 weekly from week 7-12.
2. Vinblastine IV one day a week for 6 more weeks.
3. Methotrexate given as a 24 hour IV infusion day 1 of week 7, 9, and 11, followed by leucovorin.

   * If the disease is gone or better after this additional therapy continuation will begin.

Continuation Therapy:

1. 6-MP by mouth daily until the end of month 12.
2. Prednisone in 3 doses daily days 1-5 every 3 weeks until the end of month 12.
3. Vinblastine IV day 1 every 3 weeks until the end of month 12.
4. Methotrexate by mouth once weekly until the end of month 12.

Those patients whose disease didn't respond to the initial research program by the 12th week will come off this research study and proceed to another research program.

ELIGIBILITY:
Inclusion Criteria:

All newly diagnosed patients who meet the following criteria are eligible to be enrolled and followed in the study:

* Definitive diagnosis of LCH
* Age under 18 years
* No prior treatment for LCH

Exclusion Criteria:

* Not specified

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
The proportion of non-responder in risk organs to the initial treatment | 12 months

SECONDARY OUTCOMES:
Overall survival | 12 months
Proportion of responders (overall and in risk organs) | at week 6
Proportion of responders (overall and in risk organs) | at week 12
Reactivation free survival after response | at week 12
Time to NAD | at weeks 6, 12, 7, or 13-23

CONTACTS AND LOCATIONS:
Overall Officials: Jami Frost, M.D., Principal Investigator — University of New Mexico
Locations (1):
- University of New Mexico, Albuquerque, New Mexico, United States